CLINICAL TRIAL: NCT02756182
Title: Comparison of Air-filled and Water-filled Catheters for Use in Cystometric Assessment
Brief Title: Air-charged vs Water-filled Catheters (Bonn)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AvW-Bonn-01
Record Dates: First submitted 2016-04-19; First posted 2016-04-29 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Urodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urodynamics with AC and WP (Experimental): Patients underwent a conventional urodynamics study utilizing a single catheter technique
  Interventions: Device: TDOC air-charged catheter

INTERVENTIONS:
Device: TDOC air-charged catheter — Urodynamic study utilizing a single catheter technique to measure WP & AC measurements

SUMMARY:
A comparative study was conducted and the patient underwent a conventional urodynamic study. In order to successfully determine if the Air-Charged (AC) and Water-Perfused (WP) measurements are equivalent, the two sources of intravesical pressure (Pves) and abdominal pressure (Pabd) were collected concurrently at various fill volumes for the bladder.

DETAILED DESCRIPTION:
The objective of this study was to compare the use of water-filled and air-charged catheters in determining equivalency between the two technologies during cystometric assessment.

A total of 25 patients (9M/16F) were recruited. All patients underwent cough and Valsalva manoeuvre pressure tests to measure vesicle pressure (Pves) and abdominal pressure (Pabd). A single dual-lumen catheter (T-DOC 7Fr Air-Charged® catheter) was used to record air and water pressures simultaneously.

The primary outcome was to determine if the maximum pressures during Valsalva manoeuvres, as measured with a single dual-lumen water-perfused and air-charged catheter, are equivalent when the bladder is filled to 200 cc during a urodynamic evaluation.

Exploratory endpoints included the following:

1. To determine if maximum pressures for cough, as measured with a single dual-lumen water-perfused and air-charged catheter, are equivalent when the bladder is filled to 100, 200 and Maximum Bladder Capacity (MBC) cc during a urodynamic evaluation.
2. To determine if maximum pressures for Valsalva manoeuvres, as measured with a single dual-lumen water-perfused and air-charged catheter, are equivalent when the bladder is filled to 100 and MBC cc during a urodynamic evaluation (as well as 200 cc which is the primary objective).
3. To determine if the maximum voiding pressure, as measured with a single dual-lumen water-perfused and air-charged catheter, are equivalent.
4. To determine if the clinical impressions of the urodynamic study are equivalent for the water-perfused and air-charged catheters.
5. To determine if the compliance of the bladder is equivalent when measured by air-charged catheters as compared to water-perfused catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients normally indicated for urodynamic evaluations

Exclusion Criteria:

* Patients who suffer from bladder infections (not including patients with asymptomatic bacteruria, prophylaxis with an antibiotic is at the discretion of the physician)
* Patients who suffer from strictures in the urethra
* Patients who are pregnant
* Patients who require the use of a suprapubic catheter

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Urodynamics With Air-Charged and Water Perfused: Patients underwent a conventional urodynamics study utilizing a single catheter technique
  TDOC air-charged catheter: Urodynamic study utilizing a single catheter technique to measure Water Perfused (WP) & Air-Charged (AC) measurements
Period: Overall Study
Arm/Group | Urodynamics With Air-Charged and Water Perfused
Started | 25
Completed | 21
Not Completed | 4
Not completed — StudyTechnical Difficulties | 4

BASELINE CHARACTERISTICS:
Arm/Group | Urodynamics With AC and WP
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 43.3 [21 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Vesical Pressure During Valsalva Manoeuvres
Description: Maximum vesical pressure during Valsalva manoeuvres was measured with an air-filled catheter and the water pressure was measured from the fill port. Air-filled catheter and water pressure measurements were compared.
Time Frame: Measured during a single urodynamic evaluation
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Urodynamics With AFC: Patients underwent a conventional urodynamics study utilizing a single catheter technique
  TDOC air-charged catheter: Urodynamic study utilizing a single catheter technique to measure AFC measurements
- Urodynamics With WFC: Patients underwent a conventional urodynamics study utilizing a single catheter technique
  TDOC air-charged catheter: Urodynamic study utilizing a single catheter technique to measure WFC measurements
Arm/Group | Urodynamics With AFC | Urodynamics With WFC
Number analyzed (Participants) | 21 | 21
cmH2O | 39.31 (23.02) | 39.44 (23.34)

2. Primary Outcome: Maximum Abdominal Pressure During Valsalva Manoeuvres
Description: Maximum abdominal pressure during Valsalva manoeuvres was measured with an air-filled catheter and the water pressure was measured from the fill port. Air-filled catheter and water pressure measurements were compared.
Time Frame: Measured during a single urodynamic evaluation
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Urodynamics With WFC: Patients underwent a conventional urodynamics study utilizing a single catheter technique
  Urodynamic study utilizing a single catheter technique to measure WFC measurements
Arm/Group | Urodynamics With AFC | Urodynamics With WFC
Number analyzed (Participants) | 21 | 21
cmH2O | 37.93 (21.70) | 38.11 (22.04)

3. Primary Outcome: Maximum Detrusor Pressure at Valsalva Manoeuvres
Description: Maximum detrusor pressure during Valsalva manoeuvres was measured with an air-filled catheter and the water pressure was measured from the fill port. Air-filled catheter and water pressure measurements were compared.
Time Frame: Measured during a single urodynamic evaluation
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Urodynamics With AFC | Urodynamics With WFC
Number analyzed (Participants) | 21 | 21
cmH2O | 1.72 (3.85) | 1.65 (3.39)

4. Secondary Outcome: Maximum Vesical Pressure During Coughs
Description: Maximum vesical pressure during coughs was measured with an air-filled catheter and the water pressure was measured from the fill port. Air-filled catheter and water pressure measurements were compared.
Time Frame: Measured during a single urodynamic evaluation
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Urodynamics With AFC | Urodynamics With WFC
Number analyzed (Participants) | 21 | 21
cmH2O | 64.59 (39.21) | 69.65 (43.25)

5. Secondary Outcome: Maximum Abdominal Pressure During Coughs
Description: Maximum abdominal pressure during coughs was measured with an air-filled catheter and the water pressure was measured from the fill port. Air-filled catheter and water pressure measurements were compared.
Time Frame: Measured during a single urodynamic evaluation
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Urodynamics With AFC | Urodynamics With WFC
Number analyzed (Participants) | 21 | 21
cmH2O | 60.71 (35.66) | 63.01 (38.67)

6. Secondary Outcome: Maximum Detrusor Pressure During Coughs
Description: Maximum detrusor pressure during coughs was measured with an air-filled catheter and the water pressure was measured from the fill port. Air-filled catheter and water pressure measurements were compared.
Time Frame: Measured during a single urodynamic evaluation
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Urodynamics With AFC | Urodynamics With WFC
Number analyzed (Participants) | 21 | 21
cmH2O | 3.89 (9.44) | 6.83 (7.82)

ADVERSE EVENTS:
Arm/Group | Urodynamics With AC and WP
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urodynamics With AC and WP (N=25)
High blood pressure with autonomic dysreflexia (Blood and lymphatic system disorders) | 1 (1) — One patient presented an episode of high blood pressure with autonomic dysreflexia, and the infusion pump was therefore stopped at 335 ml before maximum capacity was reached. Adverse event was not related to the device used (catheter).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No